CLINICAL TRIAL: NCT05570448
Title: Anti-Reflux Endoscopic Therapy Using Argon Plasma Coagulation (AREA) in Gastroesophageal Reflux Disease (GERD) Patients: A Single Center, Randomized, Sham, Controlled Trial (The AREA Study)
Brief Title: Anti-Reflux Endoscopic TX Using APC (AREA) in GERD Patients: (The AREA Study)
Acronym: AREA21
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Midwest Veterans' Biomedical Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PS0100; 1650419 (Other: IRBnet)
Record Dates: First submitted 2022-09-29; First posted 2022-10-06 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2022-10

CONDITIONS: Gastro Esophageal Reflux
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anti-reflux mucosal ablation (ARAT) (Active Comparator): ablation in the gastric cardia using hybrid argon plasma coagulation
  Interventions: Procedure: ARAT
- No treatment (Sham Comparator): no ablation
  Interventions: Procedure: Sham intervention (control)

INTERVENTIONS:
Procedure: ARAT — For patients randomized to ARAT intervention, the area of cardia, along greater curvature will be cleaned followed by demarcation of a 1-1.5 cm area of non-ablation zone with two vertical lines by use of Pulsed APC (30W, Effect 2) using the H-APC catheter. Next, the area of cardia, on either side will be injected in sequence using a methylene blue (0.5%) and normal saline (0.9%) using the H-APC catheter jet system (Effect 30-70). Next, the mucosa, starting below the z-line and up to 3 cm below will be treated by Pulsed APC 50W-80W till golden-brown discoloration of the ablated tissue in 270-320 degree. For patients randomized to control or sham intervention, upper endoscopy with procedural sedation was performed followed by markings of landmarks followed by gastroscope retroflexion in the gastric cardia with at least 15 minute of examination time. No H-APC or submucosal injection or other intervention will be performed.
  Other Names: Anti-reflux mucosal ablation
  Arms: Anti-reflux mucosal ablation (ARAT)
Procedure: Sham intervention (control) — Patients randomized to the control arm, will undergo a sham intervention. This will include performing upper endoscopy with procedural sedation followed by markings of landmarks as described. This will be followed by gastroscope retroflexion in the gastric cardia with at least 15 minute of examination time spent in retroflexion to reciprocate the H-APC intervention. No H-APC or submucosal injection or other intervention will be performed during the upper endoscopy with sham intervention. All Patients will also continue their PPI daily for 4 weeks.
  Arms: No treatment

SUMMARY:
This will be a randomized clinical trial examining the efficacy and safety of ARAT (intervention group) in patients with chronic GERD symptoms (typical symptoms of GERD, i.e. heartburn or acid reflux/regurgitation at least twice a week) for the last 6 months.

Patients must have a positive pH test and a negative manometry (no treatment) procedure.

ELIGIBILITY:
Inclusion Criteria:

* Chronic GERD symptoms (at least 1 typical symptom of GERD, i.e. heartburn or acid reflux/regurgitation at least twice a week) for last 6 months
* Objective evidence of reflux disease (positive ambulatory pH study.)

Exclusion Criteria:

* Patients unable to or unwilling to participate or consent.
* Age <18 years or >80 years.
* Allergic or intolerant to PPI medications.
* Large hiatal hernia > 3 cm and Hill grade IV.
* Barrett's esophagus.
* Esophageal stricture with any prior intervention.
* Major motility disorder.
* Eosinophilic esophagitis.
* Gastroparesis documented by abnormal gastric emptying time.
* Previous fundoplication, myotomy or LINX surgery.
* Cirrhosis with esophageal and/or gastric varices.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2022-02-15 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Change in GERD health related quality of life (GERD-HRQL) score | At 3, 6 and 12 months
  The primary outcome of quality of life will be measured using the validated GERD related quality of life questionnaire (GERD-HRQL). The total score is 50, and a higher score is associated with more severe symptoms.

SECONDARY OUTCOMES:
Change in Reflux disease questionnaire (RDQ) score | At 3, 6 and 12 months
  RDQ scores will be assessed using a validated questionnaire scale. The total score is 40, and a higher score is associated with more severe symptoms.
Change in Proton pump inhibitor (PPI) use | At 3, 6 and 12 months
  Frequency of PPI medication use
Acid exposure time (AET) | At 3 and 12 months
  Ambulatory acid reflux testing (wireless pH monitoring system) for measurement. Acid exposure time measures amount of time spent in pH <4. A time >4% is considered positive for acid reflux.
Adverse events | Post-randomization (Day 1, Day 30, 3rd, 6th and 12th month)
  Frequency of any adverse event including chest pain, bleeding, dysphagia, hospitalization
Change in Hiatal hernia grading | At 3 and 12 months
  Hill grade for hiatal hernia assessment during endoscopy. There are 4 grades: I, II, III and IV depending on the appearance of the hiatus on endoscopy.
Esophagitis incidence | At 3 and 12 months
  LA grade esophagitis at the time of endoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Prateek Sharma, MD, Principal Investigator — Kansas City VA Hospital; Madhav Desai, MD, Study Director — Kansas City VA Hospital
Locations (1):
- Kansas City VA Hospital, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Locke GR 3rd, Talley NJ, Fett SL, Zinsmeister AR, Melton LJ 3rd. Prevalence and clinical spectrum of gastroesophageal reflux: a population-based study in Olmsted County, Minnesota. Gastroenterology. 1997 May;112(5):1448-56. doi: 10.1016/s0016-5085(97)70025-8. PMID 9136821
- [Background] El-Serag HB, Sweet S, Winchester CC, Dent J. Update on the epidemiology of gastro-oesophageal reflux disease: a systematic review. Gut. 2014 Jun;63(6):871-80. doi: 10.1136/gutjnl-2012-304269. Epub 2013 Jul 13. PMID 23853213
- [Background] Hampel H, Abraham NS, El-Serag HB. Meta-analysis: obesity and the risk for gastroesophageal reflux disease and its complications. Ann Intern Med. 2005 Aug 2;143(3):199-211. doi: 10.7326/0003-4819-143-3-200508020-00006. PMID 16061918
- [Background] Yadlapati R, Vaezi MF, Vela MF, Spechler SJ, Shaheen NJ, Richter J, Lacy BE, Katzka D, Katz PO, Kahrilas PJ, Gyawali PC, Gerson L, Fass R, Castell DO, Craft J, Hillman L, Pandolfino JE. Management options for patients with GERD and persistent symptoms on proton pump inhibitors: recommendations from an expert panel. Am J Gastroenterol. 2018 Jul;113(7):980-986. doi: 10.1038/s41395-018-0045-4. Epub 2018 Apr 24. PMID 29686276
- [Background] Delshad SD, Almario CV, Chey WD, Spiegel BMR. Prevalence of Gastroesophageal Reflux Disease and Proton Pump Inhibitor-Refractory Symptoms. Gastroenterology. 2020 Apr;158(5):1250-1261.e2. doi: 10.1053/j.gastro.2019.12.014. Epub 2019 Dec 19. PMID 31866243
- [Background] Vaezi MF, Yang YX, Howden CW. Complications of Proton Pump Inhibitor Therapy. Gastroenterology. 2017 Jul;153(1):35-48. doi: 10.1053/j.gastro.2017.04.047. Epub 2017 May 19. PMID 28528705
- [Background] Maret-Ouda J, Wahlin K, El-Serag HB, Lagergren J. Association Between Laparoscopic Antireflux Surgery and Recurrence of Gastroesophageal Reflux. JAMA. 2017 Sep 12;318(10):939-946. doi: 10.1001/jama.2017.10981. PMID 28898377
- [Background] Witteman BP, Conchillo JM, Rinsma NF, Betzel B, Peeters A, Koek GH, Stassen LP, Bouvy ND. Randomized controlled trial of transoral incisionless fundoplication vs. proton pump inhibitors for treatment of gastroesophageal reflux disease. Am J Gastroenterol. 2015 Apr;110(4):531-42. doi: 10.1038/ajg.2015.28. Epub 2015 Mar 31. PMID 25823768
- [Background] Hillman L, Yadlapati R, Whitsett M, Thuluvath AJ, Berendsen MA, Pandolfino JE. Review of antireflux procedures for proton pump inhibitor nonresponsive gastroesophageal reflux disease. Dis Esophagus. 2017 Sep 1;30(9):1-14. doi: 10.1093/dote/dox054. PMID 28859357
- [Background] Hernandez Mondragon OV, Zamarripa Mottu RA, Garcia Contreras LF, Gutierrez Aguilar RA, Solorzano Pineda OM, Blanco Velasco G, Murcio Perez E. Clinical feasibility of a new antireflux ablation therapy on gastroesophageal reflux disease (with video). Gastrointest Endosc. 2020 Dec;92(6):1190-1201. doi: 10.1016/j.gie.2020.04.046. Epub 2020 Apr 25. PMID 32343977
- [Background] Inoue H, Tanabe M, de Santiago ER, Abad MRA, Shimamura Y, Fujiyoshi Y, Ueno A, Sumi K, Tomida H, Iwaya Y, Ikeda H, Onimaru M. Anti-reflux mucosal ablation (ARMA) as a new treatment for gastroesophageal reflux refractory to proton pump inhibitors: a pilot study. Endosc Int Open. 2020 Feb;8(2):E133-E138. doi: 10.1055/a-1031-9436. Epub 2020 Jan 22. PMID 32010745
- [Background] Taieb S, Rolachon A, Cenni JC, Nancey S, Bonvoisin S, Descos L, Fournet J, Gerard JP, Flourie B. Effective use of argon plasma coagulation in the treatment of severe radiation proctitis. Dis Colon Rectum. 2001 Dec;44(12):1766-71. doi: 10.1007/BF02234452. PMID 11742159
- [Background] Sami SS, Al-Araji SA, Ragunath K. Review article: gastrointestinal angiodysplasia - pathogenesis, diagnosis and management. Aliment Pharmacol Ther. 2014 Jan;39(1):15-34. doi: 10.1111/apt.12527. Epub 2013 Oct 20. PMID 24138285
- [Background] Peerally MF, Bhandari P, Ragunath K, Barr H, Stokes C, Haidry R, Lovat L, Smart H, Harrison R, Smith K, Morris T, de Caestecker JS. Radiofrequency ablation compared with argon plasma coagulation after endoscopic resection of high-grade dysplasia or stage T1 adenocarcinoma in Barrett's esophagus: a randomized pilot study (BRIDE). Gastrointest Endosc. 2019 Apr;89(4):680-689. doi: 10.1016/j.gie.2018.07.031. Epub 2018 Aug 1. PMID 30076843
- [Background] Manner H, Neugebauer A, Scharpf M, Braun K, May A, Ell C, Fend F, Enderle MD. The tissue effect of argon-plasma coagulation with prior submucosal injection (Hybrid-APC) versus standard APC: A randomized ex-vivo study. United European Gastroenterol J. 2014 Oct;2(5):383-90. doi: 10.1177/2050640614544315. PMID 25360316
- [Background] Inoue H, Ito H, Ikeda H, Sato C, Sato H, Phalanusitthepha C, Hayee B, Eleftheriadis N, Kudo SE. Anti-reflux mucosectomy for gastroesophageal reflux disease in the absence of hiatus hernia: a pilot study. Ann Gastroenterol. 2014;27(4):346-351. PMID 25330784
- [Background] Desjardin M, Luc G, Collet D, Zerbib F. 24-hour pH-impedance monitoring on therapy to select patients with refractory reflux symptoms for antireflux surgery. A single center retrospective study. Neurogastroenterol Motil. 2016 Jan;28(1):146-52. doi: 10.1111/nmo.12715. Epub 2015 Nov 3. PMID 26526815
- [Background] Fayad L, Oberbach A, Schweitzer M, Askin F, Voltaggio L, Larman T, Enderle M, Hahn H, Khashab MA, Kalloo AN, Kumbhari V. Gastric mucosal devitalization (GMD): translation to a novel endoscopic metabolic therapy. Endosc Int Open. 2019 Dec;7(12):E1640-E1645. doi: 10.1055/a-0957-3067. Epub 2019 Nov 25. PMID 31788546
- [Result] Vakil N, van Zanten SV, Kahrilas P, Dent J, Jones R; Global Consensus Group. The Montreal definition and classification of gastroesophageal reflux disease: a global evidence-based consensus. Am J Gastroenterol. 2006 Aug;101(8):1900-20; quiz 1943. doi: 10.1111/j.1572-0241.2006.00630.x. PMID 16928254
- See also: , Kalapala R, Nabi Z, et al. Anti-Reflux Mucosal Ablation (ARMA) For Refractory Gastroesophageal Reflux Disease - An Interim Analysis, 2021. — https://www.semanticscholar.org/paper/Anti-Reflux-Mucosal-Ablation-(ARMA)-For-Refractory-Kalapala-Jagtap/744a295131bedf263ba6f4c13126d0c5afc93b14